CLINICAL TRIAL: NCT01033006
Title: Axillary Plexus Block in a High Resolution MRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Trygve Kjelstrup, MD, Section manager, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: S-04115
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Nerve Block; Magnetic Resonance Imaging
Keywords: Peripheral Nerves; Axillary Block; MRI

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: catheter injection (Active Comparator): 40 ml of LA through the catheter
  Interventions: Procedure: Active Comparator: Arm 1: catheter injection
- Arm 2: transarterial injection (Active Comparator): 30 ml deep and 10 ml superficial to the artery
  Interventions: Procedure: Active Comparator: Arm 2: transarterial injection
- Arm 3: catheter and transarterial injection (Active Comparator): 20 + 10 ml transarterial block and 10 ml through the catheter
  Interventions: Procedure: Active Comparator: Arm 3: catheter and transarterial injection

INTERVENTIONS:
Procedure: Active Comparator: Arm 1: catheter injection
  Arms: Arm 1: catheter injection
Procedure: Active Comparator: Arm 2: transarterial injection
  Arms: Arm 2: transarterial injection
Procedure: Active Comparator: Arm 3: catheter and transarterial injection
  Arms: Arm 3: catheter and transarterial injection

SUMMARY:
Background and aims:

Magnetic resonance imaging (MRI) has proved beneficial for presenting anatomy for regional anaesthesia and to demonstrate spread of local anaesthetic.

A new axillary plexus block with a triple injection (1), combining a short axillary catheter method with a transarterial axillary block, is now being evaluated with a 3 Tesla MRI. In this study, the investigators are investigating MR visualisation of three different block techniques and compare the clinical efficacy of the techniques, with the MR findings.

Patients & Methods:

After obtaining approval of the protocol from the regional ethical committee, 3 x 15 adult patients, scheduled for hand surgery, were included in a randomised, blinded prospective study.

DETAILED DESCRIPTION:
After obtaining approval of the protocol from the regional ethical committee, 3 x 15 adult patients, scheduled for hand surgery, were included in a randomised, blinded prospective study.

In all patients a short axillary plexus catheter is positioned close to the median nerve using nerve stimulator.

Technique 1 = 40 ml in catheter Technique 2 = 30 ml behind and 10 ml in front of the brachial artery (BA) Technique 3 = 20 ml behind, 10ml in front of the BA and 10 ml in catheter

Clinical High Field MRI (3T) scanner has simplified the recognition of brachial plexus nerves in the axilla. After injection of local anaesthetic (LA), the identification of the nerve structures is nevertheless difficult. When all nerves are surrounded of LA in the axilla (MRI), it seems to be associated with a clinical complete brachial plexus block

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for hand surgery
* ASA 1 - 2
* Weight from 50 - 95 kg
* MR compatible, suitable

Exclusion Criteria:

* Neurologic deficit
* Reaction to LA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-01; Primary Completion 2011-02 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy of the blocks used compared with MRI findings | One year

CONTACTS AND LOCATIONS:
Overall Officials: Trygve TK Kjelstrup, MD, Principal Investigator — Diakonhjemmet Sykehus, University of Oslo; Øivind ØK Klaastad, PhD, MD, Study Director — Rikshospitalet, Dep. of Anesthesiology, Oslo University Hospital
Locations (1):
- The Intervention Centre, Rikshospitalet, Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Kjelstrup T, Hol PK, Courivaud F, Smith HJ, Rokkum M, Klaastad O. MRI of axillary brachial plexus blocks: a randomised controlled study. Eur J Anaesthesiol. 2014 Nov;31(11):611-9. doi: 10.1097/EJA.0000000000000122. PMID 25051144
- See also: The Intervention Centre — http://ivs.no